CLINICAL TRIAL: NCT04676659
Title: Phase II Dose-finding Open Study of Recombinant Human TNK Tissue-type Plasminogen Activator (rhTNK-tPA) Injection Administered Within 3 Hours After Onset of Hyperacute Ischemic Stroke
Brief Title: Tenecteplase Reperfusion Therapy in Acute Ischemic Cerebrovascular Events(TRACE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: CSPC Mingfule Pharmaceutical (Guangzhou) Co., Ltd. (Industry); The First Hospital Of Qiqihar (Unknown); Hebei Medical University Third Hospital (Other); Yantai Yuhuangding Hospital (Other); Fudan University (Other); First Affiliated Hospital of Jinan University (Other); The First Hospital of Jilin University (Other); Huashan Hospital (Other); West China Hospital (Other); Inner Mongolia Baogang Hospital (Other); Linyi People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Baotou Central Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Vice President of Beijing Tiantan Hospital, Capital Medical University, Director of Neurology Center, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MK02-2016-01
Record Dates: First submitted 2020-07-27; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Acute Ischemic Stroke
Keywords: rhTNK-tPA; acute; stroke; phaseII; Acute Ischemic Stroke; rt-PA
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — TNK-tissue plasminogen activator

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective, randomization, open label, active and parallel control
Who Masked: Outcomes Assessor
Masking Description: open to patient, medical cares, and investigators, but blind to outcome evaluators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (rhTNK-tPA 0.10 mg/kg) (Experimental): Dissolve one vial of rhTNK-tPA in 3 ml sterile water for injection to prepare a solution of 5.33 mg/ml. Calculate the required volume according to the body weight of the subject, then measure the required volume. Administer as a single 0.10 mg/kg IV bolus over 5-10 seconds.
  Interventions: Drug: TNK-tPA
- Group 2 (rhTNK-tPA 0.25 mg/kg) (Experimental): Dissolve one vial of rhTNK-tPA in 3 ml sterile water for injection to prepare a solution of 5.33 mg/ml. Calculate the required volume according to the body weight of the subject, then measure the required volume. Administer as a single 0.25 mg/kg IV bolus over 5-10 seconds.
  Interventions: Drug: TNK-tPA
- Group 3 (rhTNK-tPA 0.32 mg/kg) (Experimental): Dissolve one vial of rhTNK-tPA in 3 ml sterile water for injection to prepare a solution of 5.33 mg/ml. Calculate the required volume according to the body weight of the subject, then measure the required volume. Administer as a single 0.32 mg/kg IV bolus over 5-10 seconds.
  Interventions: Drug: TNK-tPA
- Group 4 (rt-PA 0.9 mg/kg) (Active Comparator): 10% of rt-PA 0.9 mg/kg administered as an initial IV bolus followed by the remaining 90% as an IV infusion over the next 1 hour.
  Interventions: Drug: TNK-tPA

INTERVENTIONS:
Drug: TNK-tPA — Experimental arms for low, middle, and high dosing; and active control arm for the standard protocol
  Other Names: rtPA

SUMMARY:
To explore the safe and efficacious dose of rhTNK-tPA injection administered within 3 hours after onset of hyperacute ischemic stroke; to provide dose evidence for phase III clinical trial.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of rhTNK-tPA at different doses of 0.10 mg/kg, 0.25 mg/kg and 0.32 mg/kg compared with standard rt-PA intravenous thrombolytic therapy within 3 hours after onset of ischemic stroke. The primary objective of this study is to evaluate the differences of NIHSS scores among the four treatment groups at 14 days after intravenous thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. Time from onset to treatment < 3 hours; the time symptoms start is defined as "the last moment they appear normal".
3. Diagnosis of ischemic stroke according to "2014 China Guideline for Diagnosis and Treatment of Acute Ischemic Stroke" with assessable neurological impairment e.g., language, motor function, cognitive impairment, gaze impairment, visual field deficit and/or visual neglect. Ischemic stroke is defined as sudden acute focal neurological impairment with suspected cerebral ischemia, hemorrhage ruled out by CT scan.
4. mRS > 2 at the first onset or prior onset.
5. Baseline NIHSS score is > 4 and < 26.
6. Signed informed consent.

Exclusion Criteria:

1. Absolute contraindications:

   1.1 History of severe head trauma or stroke within 3 months; 1.2 Suspected subarachnoid hemorrhage; 1.3 Arterial puncture at a non-compressible site within the previous 1week; 1.4 History of intracranial hemorrhage; 1.5 Intracranial tumor, vascular malformation, or arterial aneurysm; 1.6 Recent intracranial or intraspinal surgery; 1.7 Systolic blood pressure ≧ 180 mm Hg, or diastolic blood pressure ≧ 100 mm Hg; Increased blood pressure; 1.8 Active internal bleeding ; 1.9 Acute bleeding tendency, including platelet count below 100×109/L or otherwise; 1.10 Heparin treatment was performed within 48 h ( APTT exceeded the upper limit of normal range ) ; 1.11 Warfarin has been taken orally , and the international standardized ratio is INR > 1.7 or PT > 15 s ; 1.12 Anticoagulant drugs such as thrombin inhibitor or Xa factor inhibitor , argatroban ( including new anticoagulants with unclear mechanism ) are currently being used , and various sensitive laboratory tests are abnormal ( such as live ) APTT , INR , Platelet count , Serpentine ECT of pulse enzyme setting time ; thrombin time TT or appropriate determination of Xa factor activity ) ; 1.13 Blood glucose < 2.7 mmol/L; 1.14 CT showed multilobular infarction ( low density > 1 / 3 cerebral hemisphere )
2. Relative contraindications : The risks and benefits of thrombolysis should be carefully considered and weighed in the following cases ( that is , although there is one or more relative contraindications , it is not absolutely impossible to thrombolysis ).

   2.1 Mild stroke or stroke with rapid improvement of symptoms; 2.2 Women in pregnancy ; 2.3 Symptoms of neurological impairment after seizures ; 2.4 There have been major surgical operations or serious injuries in the last 2 weeks; 2.5 There were gastrointestinal or urinary system bleeding in recent 3 weeks ; 2.6 History of myocardial infarction within 3 months.
3. Have been enrolled in rhTNK-tPA in pre-study or participated in other clinical trials within 3 months prior to screening.
4. Lactating women, or childbearing women who do not use effective contraception.
5. Known allergy to rhTNK-tPA and/or rt-PA or relevant excipients.
6. The researchers judged that not suitable to participate in this study or participate in this study may lead to greater risk for patients ;
7. Can not comply with the test program or follow-up requirements .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-05-12 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | 14 days
  Proportion of subjects with NIHSS 1 or at least 4 on the NIHSS score decreased from the baseline at day14.

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 90 days
  1. Proportion of subjects of excellent outcome defined as mRS (0-1) at 90 days.
  2. Ordinal distribution of mRS and change of proportion of subjects with mRS (0-2) at 90 days.
National Institutes of Health Stroke Scale (NIHSS) | 90 days
  Neurological impairment defined as change of NIHSS score at 90 days.
Barthel(BI) | 90 days
  Global function of daily living defined as BI ≥ 95 at 90 days.
EQ-5D | 90 days
  Quality of life measured by EQ-5D scale.

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage(sICH) | 36 hours
  Proportion of subjects with symptomatic intracranial hemorrhage (sICH) at 36 hours.
Death | 90 days
  Overall mortality rate at 90 days.
Asymptomatic intracranial hemorrhage | 90 days
  Proportion of patients with asymptomatic intracranial hemorrhage at 90 days.
Hemorrhage in other parts | 90 days
  The proportion of patients with other bleeding events was defined by GUSTO bleeding at 90 days.
AE/SAE | 90 days
  Proportion of patients with adverse events / severe adverse events at 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Wang, MD,ph.D, Study Director — IRB of Beijing Tiantan Hospital,Capital Medical University
Locations (24):
- China (24):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Ninth People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - ShenZhen Hospital ,Beijing University, Shenzhen, Guangdong
  - Affiliated Hosptial to GuiZhou Medical University, Guiyang, Guizhou
  - HaiNan Provincial People's Hospital, Haikou, Hainan
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Tangshan Workers' Hospital, Tangshan, Hebei
  - The First Hospital Of Qiqihar, Qiqihar, Heilongjiang
  - Luoyang First People's Hosptical, Luoyang, Henan
  - 1st Hospital Affiliated to Zhengzhou University, Zhengzhou, Henan
  - ChangSha 1st Municipal Hospital, Changsha, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Inner Mongolia BaoGang Hospital, Baotou, Inner Mongolia
  - Huai'an Second People's Hospital, Huai'an, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - Meihekou Central Hospital, Tonghua, Jilin
  - First People 's Hospital Of Shenyang, Shenyang, Liaoning
  - General Hospital of Northern War Zone , PLA, Shenyang, Liaoning
  - Linyi People's Hospital, Linyi, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - HuaShan Hospital Affiliated to FuDan University, Shanghai, Shanghai Municipality
  - ZhongShan Hospital ,FuDan University, Shanghai, Shanghai Municipality
  - SiChuan University HuaXi Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] CAST: randomised placebo-controlled trial of early aspirin use in 20,000 patients with acute ischaemic stroke. CAST (Chinese Acute Stroke Trial) Collaborative Group. Lancet. 1997 Jun 7;349(9066):1641-9. PMID 9186381
- [Result] Wang Z, Li J, Wang C, Yao X, Zhao X, Wang Y, Li H, Liu G, Wang A, Wang Y. Gender differences in 1-year clinical characteristics and outcomes after stroke: results from the China National Stroke Registry. PLoS One. 2013;8(2):e56459. doi: 10.1371/journal.pone.0056459. Epub 2013 Feb 13. PMID 23418571
- [Result] Wei JW, Heeley EL, Wang JG, Huang Y, Wong LK, Li Z, Heritier S, Arima H, Anderson CS; ChinaQUEST Investigators. Comparison of recovery patterns and prognostic indicators for ischemic and hemorrhagic stroke in China: the ChinaQUEST (QUality Evaluation of Stroke Care and Treatment) Registry study. Stroke. 2010 Sep;41(9):1877-83. doi: 10.1161/STROKEAHA.110.586909. Epub 2010 Jul 22. PMID 20651267
- [Result] Bandera E, Botteri M, Minelli C, Sutton A, Abrams KR, Latronico N. Cerebral blood flow threshold of ischemic penumbra and infarct core in acute ischemic stroke: a systematic review. Stroke. 2006 May;37(5):1334-9. doi: 10.1161/01.STR.0000217418.29609.22. Epub 2006 Mar 30. PMID 16574919
- [Result] Donnan GA, Baron JC, Ma H, Davis SM. Penumbral selection of patients for trials of acute stroke therapy. Lancet Neurol. 2009 Mar;8(3):261-9. doi: 10.1016/S1474-4422(09)70041-9. PMID 19233036
- [Result] Macleod MR, Petersson J, Norrving B, Hacke W, Dirnagl U, Wagner M, Schwab S; European Hypothermia Stroke Research Workshop. Hypothermia for Stroke: call to action 2010. Int J Stroke. 2010 Dec;5(6):489-92. doi: 10.1111/j.1747-4949.2010.00520.x. PMID 21086713
- [Result] Lees KR, Bluhmki E, von Kummer R, Brott TG, Toni D, Grotta JC, Albers GW, Kaste M, Marler JR, Hamilton SA, Tilley BC, Davis SM, Donnan GA, Hacke W; ECASS, ATLANTIS, NINDS and EPITHET rt-PA Study Group; Allen K, Mau J, Meier D, del Zoppo G, De Silva DA, Butcher KS, Parsons MW, Barber PA, Levi C, Bladin C, Byrnes G. Time to treatment with intravenous alteplase and outcome in stroke: an updated pooled analysis of ECASS, ATLANTIS, NINDS, and EPITHET trials. Lancet. 2010 May 15;375(9727):1695-703. doi: 10.1016/S0140-6736(10)60491-6. PMID 20472172
- [Result] Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D; ECASS Investigators. Thrombolysis with alteplase 3 to 4.5 hours after acute ischemic stroke. N Engl J Med. 2008 Sep 25;359(13):1317-29. doi: 10.1056/NEJMoa0804656. PMID 18815396
- [Result] Wahlgren N, Ahmed N, Davalos A, Hacke W, Millan M, Muir K, Roine RO, Toni D, Lees KR; SITS investigators. Thrombolysis with alteplase 3-4.5 h after acute ischaemic stroke (SITS-ISTR): an observational study. Lancet. 2008 Oct 11;372(9646):1303-9. doi: 10.1016/S0140-6736(08)61339-2. Epub 2008 Sep 12. PMID 18790527
- [Result] Davis SM, Donnan GA, Parsons MW, Levi C, Butcher KS, Peeters A, Barber PA, Bladin C, De Silva DA, Byrnes G, Chalk JB, Fink JN, Kimber TE, Schultz D, Hand PJ, Frayne J, Hankey G, Muir K, Gerraty R, Tress BM, Desmond PM; EPITHET investigators. Effects of alteplase beyond 3 h after stroke in the Echoplanar Imaging Thrombolytic Evaluation Trial (EPITHET): a placebo-controlled randomised trial. Lancet Neurol. 2008 Apr;7(4):299-309. doi: 10.1016/S1474-4422(08)70044-9. Epub 2008 Feb 28. PMID 18296121
- [Result] Lees GJ. Pharmacology of AMPA/kainate receptor ligands and their therapeutic potential in neurological and psychiatric disorders. Drugs. 2000 Jan;59(1):33-78. doi: 10.2165/00003495-200059010-00004. PMID 10718099
- [Result] Davydov L, Cheng JW. Tenecteplase: a review. Clin Ther. 2001 Jul;23(7):982-97; discussion 981. doi: 10.1016/s0149-2918(01)80086-2. PMID 11519775
- [Result] Huang X, Cheripelli BK, Lloyd SM, Kalladka D, Moreton FC, Siddiqui A, Ford I, Muir KW. Alteplase versus tenecteplase for thrombolysis after ischaemic stroke (ATTEST): a phase 2, randomised, open-label, blinded endpoint study. Lancet Neurol. 2015 Apr;14(4):368-76. doi: 10.1016/S1474-4422(15)70017-7. Epub 2015 Feb 26. PMID 25726502
- [Result] Haley EC Jr, Lyden PD, Johnston KC, Hemmen TM; TNK in Stroke Investigators. A pilot dose-escalation safety study of tenecteplase in acute ischemic stroke. Stroke. 2005 Mar;36(3):607-12. doi: 10.1161/01.STR.0000154872.73240.e9. Epub 2005 Feb 3. PMID 15692126
- [Result] Carlos A Monlina,Marc Ribo,Marta Rubiera,et al.TNK Induces Faster MCA Recanalization and Leads to Better Short- and Long-term Clinical Outcome Than Native tPA.The TNK-tPA Reperfusion Stroke Study.Stroke2008,39:527 Abstract141.
- [Result] Haley EC Jr, Thompson JL, Grotta JC, Lyden PD, Hemmen TG, Brown DL, Fanale C, Libman R, Kwiatkowski TG, Llinas RH, Levine SR, Johnston KC, Buchsbaum R, Levy G, Levin B; Tenecteplase in Stroke Investigators. Phase IIB/III trial of tenecteplase in acute ischemic stroke: results of a prematurely terminated randomized clinical trial. Stroke. 2010 Apr;41(4):707-11. doi: 10.1161/STROKEAHA.109.572040. Epub 2010 Feb 25. PMID 20185783
- [Result] Parsons M, Spratt N, Bivard A, Campbell B, Chung K, Miteff F, O'Brien B, Bladin C, McElduff P, Allen C, Bateman G, Donnan G, Davis S, Levi C. A randomized trial of tenecteplase versus alteplase for acute ischemic stroke. N Engl J Med. 2012 Mar 22;366(12):1099-107. doi: 10.1056/NEJMoa1109842. PMID 22435369
- [Result] Coutts SB, Dubuc V, Mandzia J, Kenney C, Demchuk AM, Smith EE, Subramaniam S, Goyal M, Patil S, Menon BK, Barber PA, Dowlatshahi D, Field T, Asdaghi N, Camden MC, Hill MD; TEMPO-1 Investigators. Tenecteplase-tissue-type plasminogen activator evaluation for minor ischemic stroke with proven occlusion. Stroke. 2015 Mar;46(3):769-74. doi: 10.1161/STROKEAHA.114.008504. Epub 2015 Feb 12. PMID 25677596
- [Derived] Li S, Pan Y, Wang Z, Liang Z, Chen H, Wang D, Sui Y, Zhao X, Wang Y, Du W, Zheng H, Wang Y. Safety and efficacy of tenecteplase versus alteplase in patients with acute ischaemic stroke (TRACE): a multicentre, randomised, open label, blinded-endpoint (PROBE) controlled phase II study. Stroke Vasc Neurol. 2022 Feb;7(1):47-53. doi: 10.1136/svn-2021-000978. Epub 2021 Aug 24. PMID 34429364